CLINICAL TRIAL: NCT03452618
Title: Predictive Factors for the Diagnosis of Early Noninvasive Ventilation Equipment in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Predictive Factors for the Diagnosis of Early Noninvasive Ventilation Equipment
Acronym: PREDAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/17/0201; 2017-A02202-51 (Other: ID-RCB)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: diagnostic criteria
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: The study compare the diagnostic's variables in patients who received NIV one year after diagnosis and those who did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with a NIV equipment (Experimental): Determination of diagnosis variables in a group of patient who benefit of the Non Invasive ventilation equipment one year after the diagnostic
  Interventions: Diagnostic Test: diagnosis variables
- patients without a NIV equipment (Active Comparator): Determination of diagnosis variables in a group of patient who not benefit of the Non Invasive ventilation equipment one year after the diagnostic
  Interventions: Diagnostic Test: diagnosis variables

INTERVENTIONS:
Diagnostic Test: diagnosis variables — The study compare the diagnostic variables in patients who received Non invasive ventilation equipment one year after diagnosis with the patient who don't need it. For the independent variables, the present study determine a threshold at the diagnosis for which an early fitting risk appears
  The diagnostic variable are :
  * Age of the patient
  * Sex
  * Presence of bulbar involvement or not
  * Time from onset of first symptoms to diagnosis of ALS
  * Score ALSFRS-R
  * Presence of another underlying respiratory pathology (COPD, asthma ...)
  * FVC measurement (Forced vital capacity)
  * PaCO2 measurement
  * Measure SNIP (Sniff nasal inspiratory pressure)
  * Measure of Pimax (Pressure inspiratory maximal)
  * Measurement of the nocturnal desaturation index (number of desaturation less than 90% per hour of sleep)

SUMMARY:
To compensate for insufficiency of diagnostic tools, the present study propose to look for the predictive factors of an early fitting by noninvasive ventilation.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is the most common motor neuron disease. The diagnosis of this diaphragmatic dysfunction in the ALS subject is done all too often on the occasion of a hospitalization for acute respiratory insufficiency, which aggravates then the prognosis of the patients.

The presence of these factors at diagnosis will allow more surveillance to detect early diaphragmatic insufficiency and establish a NIV (Non Invasive Ventilation), the only therapeutic measure definitely improving the quality of life and survival of patients. A clinical score will be established to determine the risk of early Non Invasive Ventilation (NIV) equipment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of amyotrophic lateral sclerosis just performed,
* Patient who do not have the criteria for fitting by NIV and who have a Vital capacity ≥ 70% of theoretical values

Exclusion Criteria:

* Patient under court bail/ guardianship
* Lack of consent for participation in the study
* Presence of criteria for setting up the NIV for diagnosis according to the HAS (HealthCare Analytics Summit) 2006 recommendations
* Vital capacity <70% of the theoretical values
* Patient under Continuous Positive Pressure (CPP) or NIV for a respiratory pathology other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-12-14 (Estimated); Study Completion 2022-12-14 (Estimated)

PRIMARY OUTCOMES:
Early Surgical Clinical Score | One year after diagnostic
  An Early Surgical Clinical Score will be established taking into account the independent variables correlated to diagnosis at early fitting.
  Clinical Variables :
  * Presence of bulbar involvement or not
  * Time from onset of first symptoms to diagnosis
  * Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) score : The Amyotrophic Lateral Sclerosis Functional Ra ting Scale (ALSFRS) is an instrument for evaluating the functional status of patients with Amyotrophic Lateral Sclerosis. It can be used to monitor functional change in a patient over time.
  * Presence of another underlying respiratory disease
  Functional Variables :
  * Time from onset of first symptoms to diagnosis of ALS
  * Presence of another underlying respiratory pathology
  * Forced Vital Capacity (FVC) measurement
  * PaCO2 measurement
  * Measure Sniff Nasal Inspiratory Pressure (SNIP)
  * Measurement of diaphragmatic activity on ultrasound
  * Parameters of the Polysomnography (PSG)

SECONDARY OUTCOMES:
Sensitivity, specificity, negative and positive predictive values | One year after the diagnostic
  Sensitivity, specificity, negative and positive predictive values of the diaphragmatic ultrasound (fraction of shortening and diaphragmatic stroke) compared to the SNIP test and for the values of PSG (Polysomnography) compared to SNIP test
Percentage of decrease | One year after the diagnostic
  % decrease in shortening fraction and diaphragmatic stroke between two quarterly reevaluations correlated with early fitting and % decrease in FVC, SNIP test et Pimax
Slope of FVC decline | One year after the diagnostic
  Slope of FVC decline before and after NIV implementation and slope of decline of shortening fraction and diaphragmatic stroke before and after NIV
Quality of life score | One year after the diagnostic
  Quality of life score by the Severe Respiratory Insufficiency (SRI) questionnaire :before and after implementation of the NIV The Severe Respiratory Insufficiency (SRI) Questionnaire: a specific measure of health-related quality of life in patients receiving home mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Dupuis, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No